CLINICAL TRIAL: NCT01153126
Title: Moderating the Negative Impact of Abnormal Screening Mammograms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: XPO8110/2009-1092; 5P50CA095817 (NIH)
Record Dates: First submitted 2010-06-28; First posted 2010-06-29 (Estimated); Last update posted 2014-03-03 (Estimated); Status verified 2014-02

CONDITIONS: Breast Cancer
Keywords: Diagnostic Imaging; Breast Screening; Breast Cancer; To be eligible for the study, subjects must:; Be females at least 18 years of age,; Have had their screening mammogram performed at the UW Breast Center,; Be able to read and write English at the 6th grade level (as shown by their, ability to understand the informed consent),; Have access to a computer with internet capability.
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- No Intervention: Usual Care (No Intervention): A group receiving usual care plus 5 reliable websites
- Intervention (Experimental): A group using the Comprehensive Health Enhancement Support System (CHESS.)
  Interventions: Behavioral: Comprehensive Health Enhancement Support System (CHESS.)

INTERVENTIONS:
Behavioral: Comprehensive Health Enhancement Support System (CHESS.) — Half of the participating women will be randomly assigned to usual care and half will be offered a fully CHESS.
  Arms: Intervention

SUMMARY:
This project evaluates the impact of CHESS-Mammo by assessing participants' health information competence, psychological distress, and satisfaction with their doctor as measured by previously validated survey questionnaires.

DETAILED DESCRIPTION:
The study consists of two parts. Part 1 (focus groups) interviewed 11 women in total (6 diagnosed with breast cancer and 5 diagnosed with benign breast disease) reinforced the need for online information during the breast diagnostic process. The focus group reviewed online CHESS-Mammo module and suggested minor changes to content. Part 2 (Evaluation) will enroll 130 women in study and compare one group (65 participants) who receives access to CHESS-Mammo to another group of women (65 participants) who receive an email message containing screening mammography information. Both groups in Part 2 will be evaluated for health information competence, psychological distress, and patient satisfaction with physician through questionnaires. An evaluation of the group that accesses the CHESS-Mammo website will be done. The reason for conducting part 2 of this study is to allow greater insight into the clinical application of a novel Interactive Cancer Communication Systems (CHESS-Mammo) early in the diagnostic workup of breast cancer. By doing this project, we may achieve an important new way of implementing CHESS-Mammo in the clinic.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for the study, subjects must:

* Be females at least 18 years of age,
* Have had their screening mammogram performed at the UW Breast Center,
* Be able to read and write English at the 6th grade level (as shown by their, ability to understand the informed consent),
* Have access to a computer with internet capability.

Exclusion Criteria:

Exclusion Criteria:

* Illiterate
* Homeless

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2010-05; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
This design will allow us to compare the health information competence, psychological distress, and patient satisfaction with their doctor among the two groups. | 3 weeks
  This is a randomized controlled trial in which half of the participants will receive access to CHESS-Mammo during their diagnostic workup of an abnormal screening mammogram, and the other half will receive basic information in addition to usual care. This design will allow us to compare the health information competence, psychological distress, and patient satisfaction with their doctor among the two groups.

CONTACTS AND LOCATIONS:
Locations (1):
- University of WI Comprehensive Cancer Center and UW Health Clinics, Madison, Wisconsin, United States